CLINICAL TRIAL: NCT01582308
Title: A Study to Assess and Compare the Pharmacokinetic and Pharmacodynamic Profiles for Sitagliptin, Saxagliptin and Vildagliptin in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study Comparing the Pharmacokinetic and Pharmacodynamic Profiles for Sitagliptin, Saxagliptin and Vildagliptin in Participants With Type 2 Diabetes Mellitus (T2DM) (MK-0431-142)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0431-142; 2011-005567-25 (EudraCT Number)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; saxagliptin; Vildagliptin; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Treatment Sequence 1 (Experimental): Sitagliptin 100 mg in Period 1 followed by saxagliptin 5 mg in Period 2 followed by vildagliptin 50 mg BID in Period 3 followed by placebo in Period 4 followed by vildagliptin 50 mg in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 2 (Experimental): Saxagliptin 5 mg in Period 1 followed by vildagliptin 50 mg in Period 2 followed by placebo in Period 3 followed by sitagliptin 100 mg in Period 4 followed by vildagliptin 50 mg BID in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 3 (Experimental): Vildagliptin 50 mg in Period 1 followed by vildagliptin 50 mg BID in Period 2 followed by sitagliptin 100 mg in Period 3 followed by saxagliptin 5 mg in Period 4 followed by placebo in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 4 (Experimental): Vildagliptin 50 mg BID in Period 1 followed by placebo in Period 2 followed by saxagliptin 5 mg in Period 3 followed by vildagliptin 50 mg in Period 4 followed by sitagliptin 100 mg in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 5 (Experimental): Placebo in Period 1 followed by sitagliptin 100 mg in Period 2 followed by vildagliptin 50 mg in Period 3 followed by vildagliptin 50 mg BID in Period 4 followed by saxagliptin 5 mg in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 6 (Experimental): Sitagliptin 100 mg in Period 1 followed by vildagliptin 50 mg in Period 2 followed by saxagliptin 5 mg in Period 3 followed by placebo in Period 4 followed by vildagliptin 50 mg BID in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 7 (Experimental): Saxagliptin 5 mg in Period 1 followed by vildagliptin 50 mg BID in Period 2 followed by vildagliptin 50 mg in Period 3 followed by sitagliptin 100 mg in Period 4 followed by placebo in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 8 (Experimental): Vildagliptin 50 mg in Period 1 followed by placebo in Period 2 followed by vildagliptin 50 mg BID in Period 3 followed by saxagliptin 5 mg in Period 4 followed by sitagliptin 100 mg in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 9 (Experimental): Vildagliptin 50 mg BID in Period 1 followed by sitagliptin 100 mg in Period 2 followed by placebo in Period 3 followed by vildagliptin 50 mg in Period 4 followed by saxagliptin 5 mg in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo
- Treatment Sequence 10 (Experimental): Placebo in Period 1 followed by saxagliptin 5 mg in Period 2 followed by sitagliptin 100 mg in Period 3 followed by vildagliptin 50 mg BID in Period 4 followed by vildagliptin 50 mg in Period 5
  Interventions: Drug: Sitagliptin 100 mg; Drug: Saxagliptin 5 mg; Drug: Vildagliptin 50 mg; Drug: Vildagliptin 50 mg BID; Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin 100 mg — Sitagliptin 100 mg: one sitagliptin 100 mg tablet once daily in the morning following a fast of at least approximately 8 hours on Days 1 through 5 in one out of five treatment periods.
  Other Names: Januvia™
Drug: Saxagliptin 5 mg — Saxagliptin 5 mg: one saxagliptin 5 mg tablet once daily in the morning following a fast of at least approximately 8 hours on Days 1 through 5 in one out of five treatment periods.
  Other Names: Onglyza™
Drug: Vildagliptin 50 mg — Vildagliptin 50 mg: one vildagliptin 50 mg tablet once daily in the morning following a fast of at least approximately 8 hours on Days 1 through 5 in one out of five treatment periods.
  Other Names: Galvus™
Drug: Vildagliptin 50 mg BID — Vildagliptin 50 mg BID: one vildagliptin 50 mg tablet BID (twice daily), once in the morning following a fast of at least approximately 8 hours and once in the evening on Days 1 through 5 in one out of five treatment periods.
  Other Names: Galvus™
Drug: Placebo — Placebo: one placebo for sitagliptin tablet once daily in the morning following a fast of at least approximately 8 hours on Days 1 through 5 in one out of five treatment periods.

SUMMARY:
A five-period crossover study to assess and compare the trough dipeptidyl peptidase IV (DPP-4) inhibition at 24-hours following the final morning dose for sitagliptin, saxagliptin and vildagliptin after 5 days of once daily dosing and vildagliptin after 5 days of twice daily dosing in participants with T2DM. The primary hypothesis is that following multiple daily dose administration to achieve steady-state drug concentrations, 100-mg sitagliptin will demonstrate greater DPP-4 inhibition at 24-hours after the final dose compared to 5-mg saxagliptin and 50-mg vildagliptin (once daily administration) in participants with T2DM. Each participant will receive all 5 treatments in randomized order. There will be a washout interval of at least 10 days between the last dose of study drug in one period and the first dose of study drug in the following period.

ELIGIBILITY:
Inclusion Criteria:

* female participants of reproductive potential must not be pregnant and agree to use (and/or have their partner use) two acceptable methods of birth control beginning at least 2 weeks prior to administration of the first dose of study drug until at least 2 weeks after the last administration of study drug
* has a body mass index between 18 and 43 kg/m^2 inclusive
* has a clinically confirmed diagnosis of T2DM
* is not currently receiving any oral antihyperglycemic medications and has a screening visit hemoglobin A1c (HbA1c) between 6.5% and 10% inclusive
* must not have been previously treated with a DPP-4 inhibitor or glucagon-like peptide-1 analogs within 12 weeks of prestudy visit
* has fasting plasma or serum glucose (FPG) ≤200 mg/dL (11.1 mmol/L) at screening and randomization
* is a non-smoker or has not used nicotine or nicotine-containing products for at least approximately the last 6 months
* is willing to follow the American Heart Association weight maintaining diet and exercise program or equivalent beginning 2 weeks prior to administration of first dose of study drug and throughout the study until the poststudy visit
* agrees to refrain from the consumption of grapefruit and grapefruit juice for at least 2 weeks prior to the start of the study and throughout the study
* agrees to refrain from the consumption of all fruit juices periodically throughout the study

Exclusion Criteria:

* is mentally or legally incapacitated, has significant emotional problems at the time of prestudy visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 years
* has an estimated creatinine clearance of ≤60 mL/min
* has a history of stroke, chronic seizures, or major neurological disorder
* has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases (with the exception of stable thyroid disease, T2DM and typical associated diseases such as hypertension and hyperlipidemia)
* must not have been previously treated with any regimen that includes insulin (injected or inhaled) for at least 3 months
* has a history of type 1 diabetes mellitus and/or history of ketoacidosis, or C peptide ≤0.8 ng/mL (≤0.26 nmol/L); or secondary forms of diabetes, acute metabolic diabetic complications or evidence of significant diabetic complications (i.e. retinopathy, neuropathy, nephropathy)
* has a history of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease
* is on a weight loss program and is not in the maintenance phase, or participant has been treated with a weight loss medication within 8 weeks of screening
* anticipates the use of any new medication(s), including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of study drug and throughout the study until the poststudy visit
* anticipates any change in dose of current stable medications
* has donated or lost 1 unit of blood within 4 weeks of the prestudy visit
* has had major surgery within 30 days prior to screening or has planned major surgery
* has a history of uncontrolled hypertension
* is taking a medication which is not permitted in the study to treat a co-morbid condition, including but not limited to cytochrome P450 3A4/5 inhibitors and inducers, P-glycoprotein 1 inhibitors, and human organic anion transporter 3 inhibitors
* consumes excessive amounts of alcohol, coffee, tea, cola, or other caffeinated beverage daily
* has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately the past 6 months
* is a nursing mother

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06-21 (Actual); Primary Completion 2012-12-04 (Actual); Study Completion 2012-12-14 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Tatosian DA, Guo Y, Schaeffer AK, Gaibu N, Popa S, Stoch A, Langdon RB, Kauh EA. Dipeptidyl peptidase-4 inhibition in patients with type 2 diabetes treated with saxagliptin, sitagliptin, or vildagliptin. Diabetes Ther. 2013 Dec;4(2):431-42. doi: 10.1007/s13300-013-0045-8. Epub 2013 Oct 26. PMID 24163113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each treatment sequence started with 2 participants in Period 1. In addition, there were 2 replacement participants; in treatment sequence 5, a participant who discontinued after period 1 (placebo treatment) was replaced and in treatment sequence 7, a participant who discontinued during period 1 (saxagliptin treatment) was replaced.
Pre-assignment Details: A washout period of at least 10 days occurred between each treatment period.
Period: Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 3 (Includes replacement for a participant who discontinued after period 1) | 2 | 3 (Includes replacement for a participant who discontinued during period 1) | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: 10-day Washout Following Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 10-day Washout Following Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 10-day Washout Following Period 3
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Period: 10-day Washout Following Period 4
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1
Completed | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8 | Treatment Sequence 9 | Treatment Sequence 10
Started | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1
Completed | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Inhibition of Dipeptidyl Peptidase IV (DPP-4) Activity at Trough
Description: Percent inhibition of DPP-4 activity at 24 hours after the Day 5 morning dose (i.e., at trough) was determined by analysis of blood samples collected from the study participants.
Time Frame: 24 hours following the final morning dose on Day 5
Population: All participants who had at least at least one measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent inhibition
Groups:
- Sitagliptin 100 mg: Sitagliptin 100 mg daily for 5 days
- Saxagliptin 5 mg: Saxagliptin 5 mg daily for 5 days
- Vildagliptin 50 mg: Vildagliptin 50 mg daily for 5 days
- Vildagliptin 50 mg BID: Vildagliptin 50 mg twice daily for 5 days
- Placebo: Placebo to sitagliptin daily for 5 days
Arm/Group | Sitagliptin 100 mg | Saxagliptin 5 mg | Vildagliptin 50 mg | Vildagliptin 50 mg BID | Placebo
Number analyzed (Participants) | 17 | 20 | 18 | 17 | 17
Percent inhibition | 91.73 [91.37 to 92.08] | 73.50 [66.56 to 79.00] | 28.88 [17.90 to 38.38] | 90.63 [88.93 to 92.06] | 3.49 [-0.66 to 7.48]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Saxagliptin 5 mg; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 18.24, 90% CI 2-sided [14.97 to 21.67]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Vildagliptin 50 mg; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 62.86, 90% CI 2-sided [58.21 to 67.74]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg vs Vildagliptin 50 mg BID; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p = 0.128, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 1.11, 90% CI 2-sided [-0.10 to 2.33]
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 88.24, 90% CI 2-sided [85.77 to 90.76]
Statistical Analysis 5: Comparison: Saxagliptin 5 mg vs Vildagliptin 50 mg; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 44.62, 90% CI 2-sided [34.51 to 55.23]
Statistical Analysis 6: Comparison: Saxagliptin 5 mg vs Vildagliptin 50 mg BID; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = -17.13, 90% CI 2-sided [-21.21 to -13.25]
Statistical Analysis 7: Comparison: Saxagliptin 5 mg vs Placebo; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 70.00, 90% CI 2-sided [58.46 to 82.20]
Statistical Analysis 8: Comparison: Vildagliptin 50 mg vs Vildagliptin 50 mg BID; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = -61.75, 90% CI 2-sided [-68.76 to -55.18]
Statistical Analysis 9: Comparison: Vildagliptin 50 mg vs Placebo; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 25.38, 90% CI 2-sided [15.37 to 35.48]
Statistical Analysis 10: Comparison: Vildagliptin 50 mg BID vs Placebo; Analysis model included fixed effects terms for treatment and period; Test type: Superiority or Other; p < .001, Linear mixed effects model — P-value of between-treatment comparison of percent inhibition of DPP-4 activity; Least squares mean difference = 87.13, 90% CI 2-sided [80.06 to 94.61]

2. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Curve 0-24 Hours (AUC 0-24hr)
Description: AUC 0-24hr is the area under the plasma drug concentration-time curve calculated for the 24 hour interval after the Day 5 morning dose.
Time Frame: Predose (0 Hours) and 0.5, 1, 2, 4, 8, 12, 13 (vildagliptin 50 mg BID only), 14 (vildagliptin 50 mg BID only), 16, 20 and 24 hours after the morning dose on Day 5
Population: All participants who had at least at least one measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Sitagliptin 100 mg | Saxagliptin 5 mg | Vildagliptin 50 mg | Vildagliptin 50 mg BID
Number analyzed (Participants) | 20 | 20 | 18 | 18
nM*hr | 7070 (25.1) | 370 (25) | 3100 (27) | 6600 (26.3)

3. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Curve 0-12 Hours (AUC 0-12hr) for Vildagliptin 50 mg BID
Description: AUC 0-12hr is the area under the plasma drug concentration-time curve calculated for the 12 hour interval after the Day 5 morning dose for the vildagliptin 50 mg BID dose only.
Time Frame: Predose (0 hours) and 0.5, 1, 2, 4, 8 and 12 hours after the morning dose on Day 5
Population: All participants who had at least at least one measurement. This outcome measure is for the vildagliptin 50 mg BID dose only; therefore, results are only presented for vildagliptin 50 mg BID dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Vildagliptin 50 mg BID
Number analyzed (Participants) | 17
nM*hr | 3720 (28.9)

4. Secondary Outcome: Pharmacokinetic Analysis: Peak Plasma Drug Concentration (Cmax)
Description: Measurement of the peak plasma drug concentration following the Day 5 morning dose.
Time Frame: Predose (0 hours) and 0.5, 1, 2, 4, 8, 12, 13 (vildagliptin 50 mg BID only), 14 (vildagliptin 50 mg BID only), 16, 20, 24, 36, 48 and 96 hours after the morning dose on Day 5
Population: All participants who had at least at least one measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Sitagliptin 100 mg | Saxagliptin 5 mg | Vildagliptin 50 mg | Vildagliptin 50 mg BID
Number analyzed (Participants) | 20 | 20 | 18 | 18
nM | 724 (31.3) | 88.8 (25.2) | 586 (37) | 759 (34.7)

5. Secondary Outcome: Pharmacokinetic Analysis: Time to the Peak Plasma Drug Concentration (Tmax)
Description: Measurement of the time to the peak plasma drug concentration following the Day 5 morning dose.
Time Frame: as for outcome 4
Population: All participants who had at least at least one measurement.
Measure: Median (Full Range); unit: hr
Arm/Group | Sitagliptin 100 mg | Saxagliptin 5 mg | Vildagliptin 50 mg | Vildagliptin 50 mg BID
Number analyzed (Participants) | 20 | 20 | 18 | 18
hr | 4 [0.5 to 8] | 1 [0.5 to 2] | 1 [0.5 to 8] | 1 [0.5 to 4]

ADVERSE EVENTS:
Time Frame: Through approximately 14 days following the last dose of study drug in Period 5
Description: Of the 22 participants, 5 participants discontinued therapy and did not complete all 5 periods of the study.
Arm/Group | Sitagliptin 100 mg | Saxagliptin 5 mg | Vildagliptin 50 mg | Vildagliptin 50 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/18 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 1/20 | 4/21 | 1/18 | 1/19 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg (N=20) | Saxagliptin 5 mg (N=21) | Vildagliptin 50 mg (N=18) | Vildagliptin 50 mg BID (N=19) | Placebo (N=21)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.